CLINICAL TRIAL: NCT07381829
Title: Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Efficacy Study of the Combination Therapy With HC010 for Injection in Patients With Advanced Solid Tumors:A Multicenter, Open-Label, Dose Range-Finding and Multiple Cohort Dose Expansion Phase Ib Clinical Trial-Lung Cancer Population
Brief Title: A Phase Ib Clinical Study on the Safety and Efficacy of HC010 Combined With Chemotherapy in Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HC Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BT-HC010-102-A
Record Dates: First submitted 2025-12-09; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor Cancer
MeSH Terms: interventions — Paclitaxel; Drug Therapy; Pemetrexed; Etoposide; Carboplatin; Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HC010 + Docetaxel (Experimental): HC010 once every 3 weeks (Q3W) by intravenous drip
  Interventions: Drug: HC010; Drug: Docetaxel
- HC010 + Paclitaxel + Carboplatin/Cisplatin (Experimental): HC010 once every 3 weeks (Q3W) by intravenous drip
  Interventions: Drug: HC010; Drug: Paclitaxel (Chemotherapy); Drug: Carboplatin/Cisplatin
- HC010 + Pemetrexed + Carboplatin/Cisplatin (Experimental): HC010 once every 3 weeks (Q3W) by intravenous drip
  Interventions: Drug: HC010; Drug: Pemetrexed; Drug: Carboplatin/Cisplatin
- HC010 + Etoposide + Carboplatin/Cisplatin (Experimental): HC010 once every 3 weeks (Q3W) by intravenous drip
  Interventions: Drug: HC010; Drug: Etoposide; Drug: Carboplatin/Cisplatin

INTERVENTIONS:
Drug: HC010 — HC010 once every 3 weeks (Q3W) by intravenous drip
Drug: Paclitaxel (Chemotherapy) — the combination chemotherapy regimens are all commonly used in clinical practice
  Arms: HC010 + Paclitaxel + Carboplatin/Cisplatin
Drug: Pemetrexed — the combination chemotherapy regimens are all commonly used in clinical practice
  Arms: HC010 + Pemetrexed + Carboplatin/Cisplatin
Drug: Etoposide — the combination chemotherapy regimens are all commonly used in clinical practice
  Arms: HC010 + Etoposide + Carboplatin/Cisplatin
Drug: Carboplatin/Cisplatin — the combination chemotherapy regimens are all commonly used in clinical practice
  Arms: HC010 + Etoposide + Carboplatin/Cisplatin; HC010 + Paclitaxel + Carboplatin/Cisplatin; HC010 + Pemetrexed + Carboplatin/Cisplatin
Drug: Docetaxel — the combination chemotherapy regimens are all commonly used in clinical practice
  Arms: HC010 + Docetaxel

SUMMARY:
Phase Ib study to evaluate the tolerability, safety, pharmacokinetics and preliminary efficacy of HC010 in combination with chemotherapy regimens in patients with advanced lung cancer and determine the recommended dose for subsequent studies.

DETAILED DESCRIPTION:
This clinical trial is a multicenter, open-label, dose range-finding and multiple cohort dose expansion Phase Ib Clinical Trial-Lung Cancer Population.The goal of this study is to evaluate the tolerability, safety, pharmacokinetics and preliminary efficacy of HC010 in combination with chemotherapy regimens in patients with advanced lung cancer and determine the recommended dose for subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

* 1. Fully understand this trial and voluntarily sign the informed consent form.
* 2. For locally recurrent or metastatic non-resectable advanced solid tumors that are diagnosed by histological or cytopathological pathology and cannot be radically treated with radiotherapy, the range-finding stage does not limit specific tumor types and previous treatment conditions, while the dose-expansion stage is limited to NSCLC without standard of care, NSCLC with EGFR-sensitive mutations and progressing after adequate EGFR-TKI therapy. First-line population with driver gene negative non-small cell lung cancer and first-line population with extensive small cell lung cancer.
* 3. At least one measurable lesion according to RECIST v1.1 (patients with only brain lesion as target lesion are not accepted).
* 4. Eastern Cancer Assistance Group (ECOG) in the United States had a performance score of 0 or 1 and did not worsen within 2 weeks prior to the first dose.
* 5. The expected survival time is more than 3 months.
* 6. Adequate organ and bone marrow function.
* 7. Females of childbearing potential must have a negative blood pregnancy test within 7 days prior to the first dose of the investigational drug and be non-lactating; Eligible patients of childbearing potential (male and female) must agree to use a reliable method of contraception (hormonal or barrier method or abstinence) with their partner for at least 6 months from signing informed consent until after the last dose of study drug. Women of non-childbearing potential may not undergo pregnancy test and contraception (postmenopausal for at least 1 year or surgically sterilized).

Exclusion Criteria:

* 1. Imaging shows that the tumor invades great vessels or is not clearly demarcated from blood vessels.
* 2. Combination of brain metastasis, meningeal metastasis and spinal cord compression.
* 3. Prior concurrent anti-programmed death receptor 1 (PD-1)/programmed death ligand (PD-L1), anti-cytotoxic T lymphocyte antigen 4 (CTLA-4), and anti-vascular endothelial growth factor (VEGF) target drugs.
* 4. Anti-tumor therapy such as radiotherapy, biological therapy, endocrine therapy, targeted therapy and immunotherapy within 4 weeks prior to the first dose of study drug.
* 5. Concomitant diseases or conditions that may significantly affect the autoimmune status, such as known or suspected active autoimmune system disease, congenital or acquired immunodeficiency, hematopoietic stem cell transplantation or organ transplantation (except keratoplasty), use of live vaccine or attenuated live vaccine within 4 weeks, and use of systemic corticosteroids and immunomodulatory drugs within 2 weeks.
* 6. Concurrent with severe, uncontrolled and unrecovered acute and chronic diseases, such as acute coronary syndrome, uncontrolled hypertension, serious or poorly controlled diabetes, interstitial pneumonia requiring hormone therapy, severe bleeding tendency or coagulation disorders within the first 6 months.
* 7. Subjects with other malignant tumors within 5 years before the first dose of study drug.
* 8. Subjects who have undergone major organ surgery (excluding aspiration biopsy) within 4 weeks prior to the first dose of study drug, or have experienced significant trauma, or require elective surgery during the trial.
* 9. Adverse reactions from previous anti-tumor treatment have not recovered to NCI-CTCAE Grade 5.0 or below.
* 10. Subjects with known hypersensitivity to other monoclonal antibodies and allergies to any preparation component of the investigational drug to be used.
* 11. Subjects with known or suspected immune-related toxicity requiring permanent discontinuation after receiving any previous immunocheckpoint inhibitor therapy.
* 12. Patients who have received prior anti-angiogenic therapy and experienced Grade ≥3 toxicity associated with anti-angiogenic therapy.
* 13. The investigator believes that the subject is not suitable to participate in this clinical study for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | From first dose to 21 days

SECONDARY OUTCOMES:
Objective response rate (ORR) as assessed by the investigator according to RECIST 1.1 criteria; | Up to approximately 2 years
Disease control rate (DCR) as assessed by the investigator according to RECIST 1.1 criteria | Up to approximately 2 years
Maximum concentration (Cmax) of HC010 | Up to approximately 2 years
Number of positive cases of HC010 anti-drug antibody (ADA) | Up to approximately 2 years
Area under the curve (AUC) of HC010 | Up to approximately 2 years
Number of participants with adverse events (AEs) | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No